CLINICAL TRIAL: NCT01338974
Title: Proteomic Signature Associated With Clinical Response to Cytarabine Based Induction Therapy in Patients With AML 56 Years and Older
Brief Title: S9031-S9333-S0112-S0301-A Biomarkers Associated With Response to Cytarabine in Samples From Older Patients With Acute Myeloid Leukemia
Status: Completed | Type: Observational
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: S9031-S9333-S0112-S0301-A; S9031-S9333-S0112-S0301-A (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2011-04-19; First posted 2011-04-20 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Leukemia
Keywords: adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with del(5q); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); recurrent adult acute myeloid leukemia; untreated adult acute myeloid leukemia; adult acute minimally differentiated myeloid leukemia (M0); adult acute myeloblastic leukemia without maturation (M1); adult acute myeloblastic leukemia with maturation (M2); adult acute myelomonocytic leukemia (M4); adult acute monoblastic leukemia (M5a); adult acute monocytic leukemia (M5b); adult erythroleukemia (M6a); adult pure erythroid leukemia (M6b); adult acute megakaryoblastic leukemia (M7)
MeSH Terms: conditions — Leukemia; Congenital Abnormalities; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Acute; Leukemia, Monocytic, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Megakaryoblastic, Acute | interventions — Gene Expression Profiling; Flow Cytometry

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: gene expression analysis
Genetic: proteomic profiling
Other: flow cytometry
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of blood and tissue from patients with cancer treated with cytarabine in the laboratory may help doctors learn more about the effects of cytarabine on cells. It may also help doctors understand how well patients respond to treatment.

PURPOSE: This research trial studies biomarkers associated with response to cytarabine in samples from older patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Refinement and testing of a multiparameter flow cytometry-based cell-signaling signature (FC classifier) associated with in vivo likelihood of complete response (CR) to cytarabine-based induction chemotherapy in elderly patients (56 years and older) newly diagnosed with non-M3 acute myeloid leukemia (AML).
* Identification of cell-signaling signature(s) associated with continuous CR to cytarabine-based induction chemotherapy at one year (CCR1) in adult patients 56 years and older with a newly diagnosed non-M3 AML.
* Identification of cell-signaling signature(s) associated with relapse-free survival at one year (RFS1) in adult patients 56 years and older with a newly diagnosed non-M3 AML who received cytarabine-based induction chemotherapy and achieved CR.
* To investigate changes in cell-signaling signature(s) between matched pre- and post-treatment specimens of relapsed/refractory patients.

OUTLINE: This is a multicenter study.

Cryopreserved specimens are incubated with cytokines (e.g., interleukins), growth factors (e.g., sargramostim or filgrastim), and chemotherapeutic agent (e.g., cytarabine, etoposide) and other modulators. Cells are then fixed, permeabilized, and stained with antibodies that recognize extracellular markers (for example, surface phenotypic markers such as clusters of differentiation, drug transporters, and receptors) in conjunction with intracellular activation-state-specific epitopes of designated signaling molecules. Subsequently, cell are analyzed by phospho-flow cytometry (FC) in a random manner (without knowledge of clinical variables and outcomes) to a training set (complete pre-specified FC) versus a testing set. Cells are also analyzed by proteomic assays. Results are then compared with individual patient scores, including predicted clinical outcomes.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed with non-M3 acute myeloid leukemia (AML)
* Pretreatment and relapse/refractory cryopreserved marrow and circulating mononuclear cells (MC) from patients who meet the following criteria:

  * Eligible and evaluable patients on study SWOG-9031, SWOG-9333 (Ara-C/DNR induction arm only), SWOG-S0112, or SWOG-S0301
  * Did not refuse consent for this use of specimens
  * Have 2+ vials of pretreatment marrow cells and/or 2+ vials of pretreatment peripheral blood cells in the Southwest Oncology Group (SWOG) AML/MDS Repository

PATIENT CHARACTERISTICS:

* See Disease Characteristics

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 56 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients enrolled on S9031, S9333, S0112 or S0301 consenting to use of specimens for future research
Sampling Method: Non-Probability Sample
Enrollment: 290 (Actual)
Dates: Start 2011-03; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Response to induction chemotherapy: complete response (CR) vs non-complete response (NR) | 1 year

SECONDARY OUTCOMES:
Complete continuous response at one year (CCR1) | 1 year
Relapse-free survival at one year (RFS1) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Radich, MD, Principal Investigator — Fred Hutchinson Cancer Center

REFERENCES:
- [Derived] Medeiros BC, Othus M, Fang M, Appelbaum FR, Erba HP. Cytogenetic heterogeneity negatively impacts outcomes in patients with acute myeloid leukemia. Haematologica. 2015 Mar;100(3):331-5. doi: 10.3324/haematol.2014.117267. Epub 2014 Dec 19. PMID 25527568
- [Derived] Medeiros BC, Othus M, Estey EH, Fang M, Appelbaum FR. Unsuccessful diagnostic cytogenetic analysis is a poor prognostic feature in acute myeloid leukaemia. Br J Haematol. 2014 Jan;164(2):245-50. doi: 10.1111/bjh.12625. Epub 2013 Oct 28. PMID 24383844